CLINICAL TRIAL: NCT03405532
Title: The Effect of the CPB on Kidney Blood Flow, Function and Oxygen Uptake During Open Heart Surgery in Patients With Diabetes Mellitus
Brief Title: Kidney Function in Diabetics During CPB (Cardio Pulmonary Bypass)
Acronym: DM-ECC
Status: Suspended | Type: Observational
Why Stopped: Not enough eligible patients leading to slow recruitment
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Maria Tholén, Principal investigator, Sahlgrenska University Hospital
Other Study IDs: SahlgrenskaUHMT02
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Kidney, CPB
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: DM-ECC — Diabetes mellitus CPB

SUMMARY:
Filtration of urine in the kidney requires sufficient oxygen supply. The filtration of urine is greater in patents with diabetes. Our theory is that the diabetic kidney has a higher oxygen demand than the non diabetic kidney thereby making the diabetic kidney more sensitive to decreased oxygen delivery following reduced blood flow. With a catheter inserted into the kidney vein we will monitor the blood flow and oxygen saturation before and during CPB, in patient with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus
* Serum creatinine < 150 micromol/L preoperative
* Heart surgery requiring CPB
* LV (left ventricle) EF >40 %
* Normal hemoglobin

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with diabetes mellitus undergoing surgery requiring CBP.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-01-11 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Renal O2 extraction | 2 years
  Renal O2 extraction measured by sampling blood from a catheter inserted into the kidney vein.

SECONDARY OUTCOMES:
GFR | 2 years
  GFR (Glomerular filtration rate), measured with CrEDTA- and PAH- clearance.
Renal blood flow | 2 years
  Change in renal blood flow measured by sampling blood from a catheter inserted into the kidney vein

CONTACTS AND LOCATIONS:
Overall Officials: Sven-Erik Ricksten, Prof, Principal Investigator — Sahlgrenska Universitetssjukhuset
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No